CLINICAL TRIAL: NCT04586712
Title: Efficacy of a Controlled Short-term Trial of Cannabidiol (CBD) Ingestion on Reducing Symptomatic Response and Facilitating Recovery After Induced Muscle Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Consortium for Medical Marijuana Clinical Outcomes Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB201903330
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Muscle Injury; Recovery; Pain Relief

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active CBD-extract (Experimental): Active Dose (2000mg/30mL hemp extract = 67.5mg/day)
  Interventions: Drug: Active CBD
- Vehicle-Control (Placebo) (Placebo Comparator): (0mg/30mL hemp extract = no hemp extract)
  Interventions: Drug: Vehicle Control (Placebo)

INTERVENTIONS:
Drug: Active CBD — Participants will be provided a viscous liquid in a bottle with a syringe dropper containing CBD-extract oil at concentrations of 2000mg/30mL (high).
  Other Names: 2000mg/30mL
  Arms: Active CBD-extract
Drug: Vehicle Control (Placebo) — Participants will be provided a viscous liquid in a bottle with a syringe dropper containing placebo containing no CBD oil (0mg/30 mL).
  Arms: Vehicle-Control (Placebo)

SUMMARY:
We aim to determine the efficacy of a controlled short-term trial of CBD ingestion for reducing symptomatic response and facilitating recovery following induced muscle injury. We will assess, in serial fashion, symptomatic response, functional limitations and recovery of the quadriceps muscle following induced injury in which CBD oil (or placebo) will be delivered using a sublingual route of administration during a 15-day pre-injury consumption and post-injury recovery phase. A double-blind, randomized, two-arm study design will be used and participants will be randomly assigned to either an active dose (n=15) or vehicle control group (n=15). The clinical outcomes include measures of muscular pain and disability along with measures of pain-related fear and anxiety.

DETAILED DESCRIPTION:
Current research has shown evidence that phytocannabinoids may have a promising therapeutic potential in a variety of physical and psychological ailments, and cannabidiol (CBD) is of particular interest due to its positive safety profile, non-intoxicating effects and widespread capabilities in a number of musculoskeletal diseases. Three primary reasons people consume CBD on a global basis, in addition to the fact that it is non-intoxicating, are for symptomatic (pain) relief, anxiety reduction, and improved sleep quality. Very little is known about CBD and how it functions in the body from both an efficacy and mechanistic perspective, especially in humans. There is a large consumer base for this product that will be expanding exponentially in the next few years. Most of the evidence available is anecdotal from the personal testimony of consumers. We aim to determine the efficacy of a controlled short-term trial of CBD ingestion for reducing symptomatic response and facilitating recovery following induced muscle injury. We will assess, in serial fashion, symptomatic response, functional limitations and recovery of the quadriceps muscle following induced injury in which selected doses of CBD oil (or placebo) will be delivered using a sublingual route of administration during a 15-day pre-injury consumption and post-injury recovery phase. A double-blind, randomized, two-arm study design will be used and participants will be randomly assigned to either an active dose (n=15) or vehicle control group (n=15). Our clinical outcomes include measures of muscular pain and disability along with measures of pain-related fear and anxiety. Our laboratory-based study design is desirable and advantageous because it is a controlled method of tracking individuals using an experimental model of injury that is translatable to clinical populations. This exploratory study will provide preliminary data needed to support the hypotheses of a planned larger scale application.

ELIGIBILITY:
Inclusion Criteria: a) male and female adults between the ages of 18-35 years and b) English speaking, and c) both female and male subjects must be currently practicing acceptable methods of birth control, such as abstinence, and methods of contraception (barriers, oral, patch or other prophylactic methods).

Exclusion Criteria: a) current use of cannabis products on a regular basis or positive urine test for cannabis, b) current use of tobacco or nicotine containing products on a regular basis, c) currently taking prescription medication for management of anxiety disorders, depression, or ADHD, d) current use of nutritional or dietary supplements on a daily basis (e.g. ephedra, yohimbine, pro-hormones, creatine or anabolics), e) current use of OTC anti-inflammatory medications (e.g. Advil, Aleve, Aspirin) on a regular basis, f) history of seizure disorder, family history of seizure disorder, current or history of head trauma, liver disease, renal (kidney) disease, cardiovascular disease (including, but not limited to: hypotension, hypertension, tachycardia, and syncope), g) current medical condition that would prevent the participant from performing strenuous resistance exercise, h) weight lifting for the lower extremities (legs) more than twice a week, i) currently experiencing pain in the hips, leg, or knee region, j) pregnancy, lactating or positive urine pregnancy test, k) known allergy to CBD or coconut/sesame oil, l) an allergy to tree nuts (coconut).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Borsa, PhD, ATC, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Started | 17 | 17
Completed | 15 | 14
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo) | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 29
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.1 (1.4) | 19.8 (1.6) | 20.0 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 12 | 13 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 9 | 17
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Self-report Ratings of Muscle Soreness
Description: A muscle soreness inventory will be used to self-report the level of soreness. The muscle soreness inventory consists of rating soreness on a visual analog scale (VAS). A 10cm line is drawn with 0 (no soreness) on the left pole and 10 (extreme soreness) on the right pole.
Time Frame: Baseline (Day 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 15 | 13
score on a scale | 0.0 (0) | 0.0 (0)

2. Primary Outcome: Self-report Ratings of Muscle Soreness
Description: as for outcome 1
Time Frame: Pre-exercise (Day 10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 15 | 13
score on a scale | 4.0 (7.4) | 2.3 (5.9)

3. Primary Outcome: Self-report Ratings of Muscle Soreness
Description: A muscle soreness inventory will be used to self-report the level of soreness. The muscle soreness inventory consists of rating soreness on a visual analog scale (VAS). A 100mm line is drawn with 0 (no soreness) on the left pole and 100 (extreme soreness) on the right pole.
Time Frame: Post-exercise (Day 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 15 | 13
score on a scale | 47.8 (27.3) | 61.6 (22.3)

4. Primary Outcome: Self-report Ratings of Disability
Description: Disability will be measured using the Lower Extremity Functional Scale (LEFS). LEFS score = SUM (points for all 20 activities) Interpretation: Minimum score: 0 Maximum score: 80 The lower the score the greater the disability.
Time Frame: Baseline (Day 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 15 | 15
score on a scale | 77.2 (5.4) | 76.7 (4.6)

5. Primary Outcome: Self-report Ratings of Disability
Description: as for outcome 4
Time Frame: Pre-exercise (Day 10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 15 | 15
score on a scale | 77.1 (4.8) | 75.9 (5.4)

6. Primary Outcome: Self-report Ratings of Disability
Description: as for outcome 4
Time Frame: Post-exercise (Day 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 15 | 15
score on a scale | 67.7 (13.2) | 60.1 (27.4)

7. Secondary Outcome: Pain Anxiety Symptom Scale - 20 (PASS-20)
Description: 20 item, 5-point rating scale that assesses 4 theoretically distinct components of pain-related anxiety including cognitive anxiety (items 1 to 5), fear of pain (items 6 to 10), escape/avoidance behavior (items 11 to 15), and physiological anxiety (items 16 to 20). Each subscale is worth 20 points. Subscales are combined to compute total score. The total scale ranges from 0 to 100; higher scores indicate worse outcome.
Time Frame: Pre-exercise (Day 10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 15 | 13
score on a scale | 39.5 (15.4) | 49.9 (22.1)

8. Secondary Outcome: Pain Anxiety Symptom Scale (PASS-20)
Description: as for outcome 7
Time Frame: Post-exercise (Day 15)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 15 | 13
score on a scale | 39.1 (16.9) | 47.9 (21.4)

9. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: 13-item, 5-point rating scale used to assess different thoughts that may be associated with experiencing pain. The PCS total score is computed by summing responses to all 13 items.
  PCS total scores range from 0 - 52. The PCS subscales are computed by summing the responses to the following items: Rumination: Sum of items 8, 9, 10, 11; Magnification: Sum of items 6, 7, 13; and Helplessness: Sum of items 1, 2, 3, 4, 5, 12; higher scores indicate worse outcome.
Time Frame: Baseline (Day 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 15 | 13
score on a scale | 21.1 (6.5) | 26.4 (11.7)

10. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: as for outcome 9
Time Frame: Pre-exercise (Day 10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 15 | 13
score on a scale | 21.3 (7.5) | 25.4 (11.2)

11. Secondary Outcome: Pain Catastrophizing Scale (PCS)
Description: as for outcome 9
Time Frame: Post-exercise (Day 15)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 15 | 13
score on a scale | 21.4 (10.1) | 23.9 (10.3)

12. Secondary Outcome: Fear of Pain Questionnaire (FPQ-9)
Description: 9-item, 5-point rating scale to quantify fear of specific situations that normally produce pain. Each subscale contains 3 items, so the possible range of scores for each subscale is 3 through 15. Subscales are combined to compute total score. The Total score has a range of 9 through 45; higher scores indicate worse outcome.
Time Frame: Baseline (Day 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 15 | 13
score on a scale | 23.8 (5.4) | 21.3 (5.7)

13. Secondary Outcome: Fear of Pain Questionnaire (FPQ-9)
Description: as for outcome 12
Time Frame: Pre-exercise (Day 10)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 15 | 13
score on a scale | 21.5 (5.0) | 18.8 (7.1)

14. Secondary Outcome: Maximal Voluntary Isometric Contraction (MVIC)
Description: maximum voluntary force produced during a static muscle contraction
Time Frame: Pre-exercise (Day 10)
Measure: Mean (Standard Deviation); unit: Newton-meters
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 13 | 12
Newton-meters | 138.5 (23.3) | 129.3 (42.1)

15. Secondary Outcome: Maximal Voluntary Isometric Contraction (MVIC)
Description: maximum voluntary force produced during a static muscle contraction measured in Newton-meters.
Time Frame: Post-exercise (Day 12)
Measure: Mean (Standard Deviation); unit: force output in Newton-meters
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 13 | 12
force output in Newton-meters | 122.4 (41.2) | 102.4 (32.6)

16. Secondary Outcome: Maximal Voluntary Isometric Contraction (MVIC)
Description: maximum voluntary force produced during a static muscle contraction measured as Newton-meters.
Time Frame: Post-exercise (Day 15)
Measure: Mean (Standard Deviation); unit: force output in Newton-meters
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
Number analyzed (Participants) | 13 | 12
force output in Newton-meters | 128.4 (50.2) | 121.0 (44.7)

ADVERSE EVENTS:
Time Frame: 15 days
Description: Self-reported by participant
Arm/Group | Active CBD-extract | Vehicle-Control (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/12/NCT04586712/Prot_SAP_001.pdf